CLINICAL TRIAL: NCT06195644
Title: Effect of Galvanic Vestibular Stimulation on Cortical Excitability and Hand Dexterity in Multiple Sclerosis Patients
Acronym: GVS on MS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hassanin, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004742
Record Dates: First submitted 2023-12-11; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Cortical Excitability; Multiple Sclerosis
Keywords: Galvanic Vestibular Stimulation; Hand Dexterity; Multiple Sclerosis; Transcranial magnetic Stimulation; Cortical excitability
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GVS group (Experimental): Galvanic Vestibular Stimulation in addition to the Conventional Physical Therapy program of moderate intensity aerobic training on cyclic ergometer for upper limb and task oriented training for hand dexterity.
  Interventions: Device: Galvanic vestibular stimulation; Device: MovAlyzeR® software from Neuroscript; Device: BODYFIT Mini Portable Pedal Home Exerciser (cyclic ergometer)
- CPT group (Active Comparator): Conventional Physical Therapy program of moderate intensity aerobic training on cyclic ergometer for upper limb and task oriented training for hand dexterity.
  Interventions: Device: MovAlyzeR® software from Neuroscript; Device: BODYFIT Mini Portable Pedal Home Exerciser (cyclic ergometer)

INTERVENTIONS:
Device: Galvanic vestibular stimulation — galvanic current generated by Gymna DUO 200 and delivered through conductive medium (electrode gel) by two small carbon rubber electrodes 3 cm 2 each bilaterally over two mastoid processes for 30 minutes, two times per week for 12 weeks .
  Arms: GVS group
Device: MovAlyzeR® software from Neuroscript — MovAlyzeR® movement analysis software from Neuroscript turns a pen tablet or mouse into a high-quality system for examining movements by a pen, mouse or finger. Hence, it can train and analyze hand dexterity and handwriting using pen tablets such as sentence parameters.
Device: BODYFIT Mini Portable Pedal Home Exerciser (cyclic ergometer) — stationary upper body pedaling as a moderate intensity aerobic training

SUMMARY:
This study will be conducted to investigate the following:

1. The impact of implementing GVS in MS rehabilitation on cortical excitability.
2. The influence of GVS on upper limb function in patients diagnosed with MS. Patients will be randomly assigned to a control group (Conventional Physical Therapy program = CPT) and a study group (Galvanic Vestibular Stimulation = GVS in addition to the conventional program) subsequently. CPT will perform moderate intensity aerobic training (arm ergometer) and task oriented hand manipulation training, while GVS will receive Galvanic Vestibular Stimulation will be added to the conventional physical Therapy program.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ataxic RRMS type of both genders will be recruited. The last MS relapse occurred at least 3 months prior to the study.
2. Patients' age will range from 20 to 45 years old.
3. Ambulant Patients who meet the level less than or equal to 5 on EDSS will be recruited.
4. Patients' score on Mini Mental State Examination should be > 26.
5. Mild or no spasticity (grade 1 or 1+) according to Modified Ashworth Scale.
6. All patients must at least hold Primary stage certificate of education from one of the Egyptian educational authorities.
7. All patients can independently sign consent form

Exclusion Criteria:

* Patients will be excluded if they have:

  1. Moderate to severe auditory or visual or cognitive impairment.
  2. Coexistence of other neurological diagnoses of Central or Peripheral Nervous system (e.g. cerebrovascular stroke, vestibulopathy or polyneuropathy).
  3. History of any problems that hinder conduction of aerobic training or magnetic stimulation (e.g. deep venous thrombosis, shunts and pacemakers).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cortical changes | 15 minutes
  central motor conduction time is the time taken for neural impulses to travel through the central nervous system on their way to the target muscles.
Upper Limb motor dexterity | 15-20 minutes
  Nine hole peg test 9 HPT

SECONDARY OUTCOMES:
Advanced dexterity (Handwriting analysis) by MovAlyzeR® software | 15-20 minutes
Balance | 15-20 minutes
  Berg Balance scale (BBS) of 14 items graded on 5 scoring system 0= worst and 4= the best ( total 0 = worst performance - Total 56 = Best performance). The lower your score, the more at risk you are for losing your balance. In general, Berg balance scale scores are interpreted as such: 0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely.
Fatigue | 15-20 minutes
  Fatigue Severity Scale (FSS)is 9-item questionnaire, scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No